CLINICAL TRIAL: NCT05199532
Title: Eosinophilic Gastrointestinal Disorders Registry
Status: Recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Joshua Wechsler, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2020-3601
Record Dates: First submitted 2021-10-06; First posted 2022-01-20 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Eosinophilic Esophagitis; Eosinophilic Gastroenteritis; Eosinophilic Colitis; Eosinophilic Gastrointestinal Disease
MeSH Terms: conditions — Eosinophilic Esophagitis; Eosinophilic enteropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — 1. Biopsies stored in AllProtect
  2. Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to learn more about Eosinophilic Gastrointestinal Disorders (EGIDs). With this registry we hope to find out more about the symptoms that patients have during their treatment, the quality of life they have with the diagnosis, what the disease looks like throughout the different treatment methods, and if there is a connection between EGIDs and connective tissue disorders.

The goal of this study is to be able to better understand EGIDs and use information gained from all the information collected on this study for more precise treatments in the future. We want to create a large collection of samples, called a biorepository, to learn the most about EGIDs as possible. When the samples are collected, which will occur at procedures directed by your child's doctor as part of their standard of care, they will be stored for an unlimited amount of time to perform experiments on these samples and to gather information about EGIDs

DETAILED DESCRIPTION:
Eosinophilic gastrointestinal disorders (EGIDs) comprise a family of disorders that includes Eosinophilic Esophagitis (EoE), Eosinophilic Gastritis (EG), Eosinophilic Gastroenteritis (EGE), and Eosinophilic Colitis (EC). The natural history of EGIDs is not well characterized. The aim of this registry is to create a comprehensive prospective database of EGID patients as a foundation towards an improved understanding of disease progression and pathophysiologic mechanism. There is a critical need to understand the relationship between disease mechanism, treatment response, measurements of disease severity, and noninvasive disease activity monitoring strategies. Characterization of the spectrum of clinical phenotype of EGIDs is important in the search for novel pathogenic molecules/pathways to inform targeted treatment strategies.

This study proposes to establish an EGID patient registry comprised of data collected from patients at Lurie Children's Hospital of Chicago undergoing standard of care evaluation, diagnosis, and treatment for EGIDs. The registry aims to characterize the clinical phenotype of EGIDs by examining (1) clinical, endoscopic, and histologic characteristics of EGID patients compared to non-EGID controls; (2) clinical, endoscopic, and histologic response of EGID patients to treatment; (3) functional assessment of the esophagus in patients undergoing evaluation for and with established diagnosis of EoE; (4) patient-reported quality of life and symptom scales; (5) the association of EGIDs with inherited Connective Tissue Disorders (CTDs) and dysautonomia, and (6) cellular and molecular biomarkers of disease severity. Our aim is to perform a prospective analysis of all EoE, EG, EGE, and EC patients, as well as patients suspected of having an EGID evaluated at Lurie Children's Hospital. Patients who are suspected of having an EGID and those with an established diagnosis of an EGID will be approached for recruitment into the registry.

The data and samples collected during this study are important to this study and to future research related to EGIDs. The data and samples will be used as indicated within this protocol and remaining samples and data will be stored and kept for future research studies on gastrointestinal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of an EGID, based on pathology findings from an endoscopy or colonoscopy with biopsies.
* Patients suspected of having an EGID and undergoing endoscopic evaluation for further assessment

Exclusion Criteria:

* Patients who do not consent to participate

Ages: 1 Year to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: The subjects of this study include patients followed at Lurie Children's Hospital for evaluation or treatment of an EGID. Patients receiving care at Lurie Children's hospital include residents of the greater Chicago area, as well as patients throughout the Midwest seeking care at a tertiary referral center. Patients suspected of having EGID present with a wide variety of symptoms, ranging from classic symptoms of EoE including dysphagia and food impaction, to more general symptoms of abdominal pain, heartburn, vomiting, food refusal, failure to thrive, and diarrhea. Diagnostic criteria for EGIDs rely on clinical symptoms and the presence of eosinophil-predominant inflammation on biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Clinical/Patient-Reported Measures | through study completion, an average of 6 months to 1 year
  Families complete questionnaires regarding reported symptoms and quality of life as well as family history, patient history and dietary checklists. Change in responses will be assessed at collection timepoints
Endoscopic measures | through study completion, an average of 6 months to 1 year
  Endoscopy visual findings will be evaluated using EREFS measurements, which measure the visual findings of Exudates, Rings, Edema, Furrows, and Strictures
Physical exam findings | through study completion, an average of 6 months to 1 year
  hypermobility as assessed by Beighton Score, assessed from 5 questions on a 0-2 scale with a higher score reporting a positive association with hypermobility
Histologic features | through study completion, an average of 6 months to 1 year
  Histology markers of eosinophilic esophagitis, specifically eos/hpf, will be assessed at standard of care endoscopies to show change throughout study participation
Molecular measures | through study completion, an average of 6 months to 1 year
  In particular, we will assess mast cells and t-cells, and their mediators that are increased in EGIDs

CONTACTS AND LOCATIONS:
Overall Officials: Joshua B Wechsler, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Dellon ES, Hirano I. Epidemiology and Natural History of Eosinophilic Esophagitis. Gastroenterology. 2018 Jan;154(2):319-332.e3. doi: 10.1053/j.gastro.2017.06.067. Epub 2017 Aug 1. PMID 28774845
- [Background] O'Shea KM, Aceves SS, Dellon ES, Gupta SK, Spergel JM, Furuta GT, Rothenberg ME. Pathophysiology of Eosinophilic Esophagitis. Gastroenterology. 2018 Jan;154(2):333-345. doi: 10.1053/j.gastro.2017.06.065. Epub 2017 Jul 27. PMID 28757265
- [Background] Jensen ET, Kappelman MD, Martin CF, Dellon ES. Health-care utilization, costs, and the burden of disease related to eosinophilic esophagitis in the United States. Am J Gastroenterol. 2015 May;110(5):626-32. doi: 10.1038/ajg.2014.316. Epub 2014 Sep 30. PMID 25267327
- [Background] Furuta GT, Katzka DA. Eosinophilic Esophagitis. N Engl J Med. 2015 Oct 22;373(17):1640-8. doi: 10.1056/NEJMra1502863. PMID 26488694
- [Background] Steinbach EC, Hernandez M, Dellon ES. Eosinophilic Esophagitis and the Eosinophilic Gastrointestinal Diseases: Approach to Diagnosis and Management. J Allergy Clin Immunol Pract. 2018 Sep-Oct;6(5):1483-1495. doi: 10.1016/j.jaip.2018.06.012. Epub 2018 Jul 3. PMID 30201096
- [Background] Dellon ES, Liacouras CA, Molina-Infante J, Furuta GT, Spergel JM, Zevit N, Spechler SJ, Attwood SE, Straumann A, Aceves SS, Alexander JA, Atkins D, Arva NC, Blanchard C, Bonis PA, Book WM, Capocelli KE, Chehade M, Cheng E, Collins MH, Davis CM, Dias JA, Di Lorenzo C, Dohil R, Dupont C, Falk GW, Ferreira CT, Fox A, Gonsalves NP, Gupta SK, Katzka DA, Kinoshita Y, Menard-Katcher C, Kodroff E, Metz DC, Miehlke S, Muir AB, Mukkada VA, Murch S, Nurko S, Ohtsuka Y, Orel R, Papadopoulou A, Peterson KA, Philpott H, Putnam PE, Richter JE, Rosen R, Rothenberg ME, Schoepfer A, Scott MM, Shah N, Sheikh J, Souza RF, Strobel MJ, Talley NJ, Vaezi MF, Vandenplas Y, Vieira MC, Walker MM, Wechsler JB, Wershil BK, Wen T, Yang GY, Hirano I, Bredenoord AJ. Updated International Consensus Diagnostic Criteria for Eosinophilic Esophagitis: Proceedings of the AGREE Conference. Gastroenterology. 2018 Oct;155(4):1022-1033.e10. doi: 10.1053/j.gastro.2018.07.009. Epub 2018 Sep 6. PMID 30009819
- [Background] Godwin B, Wilkins B, Muir AB. EoE disease monitoring: Where we are and where we are going. Ann Allergy Asthma Immunol. 2020 Mar;124(3):240-247. doi: 10.1016/j.anai.2019.12.004. Epub 2019 Dec 9. PMID 31830586
- [Background] Carlson DA, Lin Z, Hirano I, Gonsalves N, Zalewski A, Pandolfino JE. Evaluation of esophageal distensibility in eosinophilic esophagitis: an update and comparison of functional lumen imaging probe analytic methods. Neurogastroenterol Motil. 2016 Dec;28(12):1844-1853. doi: 10.1111/nmo.12888. Epub 2016 Jun 16. PMID 27311807
- [Background] Abonia JP, Wen T, Stucke EM, Grotjan T, Griffith MS, Kemme KA, Collins MH, Putnam PE, Franciosi JP, von Tiehl KF, Tinkle BT, Marsolo KA, Martin LJ, Ware SM, Rothenberg ME. High prevalence of eosinophilic esophagitis in patients with inherited connective tissue disorders. J Allergy Clin Immunol. 2013 Aug;132(2):378-86. doi: 10.1016/j.jaci.2013.02.030. Epub 2013 Apr 19. PMID 23608731
- [Background] Tinkle BT, Levy HP. Symptomatic Joint Hypermobility: The Hypermobile Type of Ehlers-Danlos Syndrome and the Hypermobility Spectrum Disorders. Med Clin North Am. 2019 Nov;103(6):1021-1033. doi: 10.1016/j.mcna.2019.08.002. PMID 31582002
- [Background] Huang KZ, Dellon ES. Increased prevalence of autonomic dysfunction due to postural orthostatic tachycardia syndrome in patients with eosinophilic gastrointestinal disorders. J Gastrointestin Liver Dis. 2019 Mar;28(1):47-51. doi: 10.15403/jgld.2014.1121.281.syd. PMID 30851172
- [Background] Fikree A, Aziz Q, Sifrim D. Mechanisms underlying reflux symptoms and dysphagia in patients with joint hypermobility syndrome, with and without postural tachycardia syndrome. Neurogastroenterol Motil. 2017 Jun;29(6). doi: 10.1111/nmo.13029. Epub 2017 Feb 12. PMID 28191707